CLINICAL TRIAL: NCT00079976
Title: A Clinical Research Study to Evaluate the Safety and Efficacy of Tigecycline in the Treatment of Selected Serious Infections Caused by Vancomycin-Resistant Enterococcus (VRE) or Methicillin-Resistant Staphylococcus Aureus (MRSA)
Brief Title: Study Evaluating Tigecycline in Selected Serious Infections Caused by Vancomycin-Resistant Enterococcus (VRE) or Methicillin-Resistant Staphylococcus Aureus (MRSA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 3074A1-307
Record Dates: First submitted 2004-03-19; First posted 2004-03-22 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Gram-Positive Bacterial Infections; Staphylococcus Infections; Vancomycin Resistance; Methicillin Resistance
Keywords: Staphylococcus aureus; Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Staphylococcal Infections; Bacterial Infections | interventions — Tigecycline

INTERVENTIONS:
Drug: Tigecycline

SUMMARY:
To evaluate the safety and efficacy of tigecycline in the treatment of selected serious infections caused by VRE. The primary efficacy endpoint will be the clinical response for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older
* Isolation of one of the following multi-antibiotic resistant bacteria: vancomycin-resistant Enterococcus faecium, vancomycin-resistant Enterococcus faecalis, or methicillin-resistant Staphylococcus aureus, alone or as part of a polymicrobial infection
* Have a confirmed diagnosis of a serious infection (eg, bacteremia [unless due to an excluded infection], complicated intra-abdominal infection, complicated skin and skin structure infection, or pneumonia) requiring administration of intravenous (IV) antibiotic therapy

Exclusion Criteria:

* Subjects with any concomitant condition or taking any concomitant medication that, in the opinion of the investigator, could preclude an evaluation of a response or make it unlikely that the contemplated course of therapy or follow-up assessment will be completed or that will substantially increase the risk associated with the subject's participation in this study
* Anticipated length of antibiotic therapy less than 7 days
* For subjects with VRE, known or suspected hypersensitivity to tigecycline or linezolid, or other compounds related to these classes of antibacterial agents (eg, oxazolidinones, tetracyclines, minocycline, doxycycline). For subjects with MRSA, known or suspected hypersensitivity to tigecycline or vancomycin, or other compounds related to these classes of antibacterial agents (eg, tetracyclines, minocycline, doxycycline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2003-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer